CLINICAL TRIAL: NCT06742021
Title: Application of DCE-MRI Based on 4D FreeBreathing in Predicting the Efficacy of Immune and Targeted Therapy in Lung Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yunnan Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KYLX2024-272
Record Dates: First submitted 2024-12-15; First posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Application Value of MRI Imaging in Treatment Decision-Making for Lung Cancer (Experimental): A Philips 3.0T MRI scanner was used, with a dStream Torso 32-channel coil. DCE-MRI was performed using a free-breathing sequence with a flow velocity of 3.0 m/s. The image quality assessment in this study was performed by two radiologists (one with 3 years of diagnostic experience and the other with 15 years of diagnostic experience), including both subjective and objective evaluations. Then, dynamic information from the 4D FreeBreathing DCE-MRI images taken before treatment and one week after immunotherapy/targeted therapy, along with routine clinical and pathological data, were used to construct predictive models for the efficacy of immunotherapy and targeted therapy. Finally, the MRI model was compared with the CT model, and the performance of both models was evaluated.
  Interventions: Diagnostic Test: Application Value of MRI Imaging in Treatment Decision-Making for Lung Cancer

INTERVENTIONS:
Diagnostic Test: Application Value of MRI Imaging in Treatment Decision-Making for Lung Cancer — Chest MRI scans outside of the standard treatment protocol

SUMMARY:
This study aims to address the challenge of predicting the efficacy of targeted and immunotherapy in lung cancer patients. By utilizing two DCE-MRI images-one before treatment and one after one treatment cycle-along with the patients' clinical and pathological information, we aim to achieve accurate prediction of the therapeutic efficacy of targeted and immunotherapy in lung cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Tumor size greater than 2 cm
2. Age between 18 and 75 years

Exclusion Criteria:

1. Presence of MRI contraindications (e.g., metal implants, pacemaker implantation, etc.)
2. Allergy to gadolinium contrast agents
3. Lesions difficult to delineate on images due to conditions such as atelectasis or diffuse lesions

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Estimated)
Dates: Start 2024-11-11 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Tumor treatment response evaluation | within one week before treatment and two weeks after treatment completion
  This study aims to evaluate tumor treatment response using the RECIST V1.1 criteria, based on CT images taken within one week before treatment and two weeks after treatment completion.

CONTACTS AND LOCATIONS:
Overall Officials: Lianhua Ye, Study Director — Ethics Committee of Yunnan Provincial Cancer Hospital
Locations (1):
- Yunnan Cancer Hospital, Kunming, Yunnan, China